CLINICAL TRIAL: NCT06333756
Title: Effects of Cross Education Training on Corticocortical and Corticomuscular Functional Connectivity
Brief Title: Effects of Muscle Strengthening and Fatigue on Activities in Cortex and Muscle
Acronym: YM110099E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: YM110099E
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2022-12

CONDITIONS: Healthy Adults
Keywords: cross education, functional connectivity

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cross education training group (Experimental): Cross education on elbow flexor
  Interventions: Other: Cross education

INTERVENTIONS:
Other: Cross education — Cross education training of the biceps brachii (12 rep./set, 3sets, 60%MVIC,180°/s, eccentric contraction)

SUMMARY:
We will explored the effect of cross education training on different cortex functional connectivity, cortex and muscle functional connectivity, and maximal voluntary contraction.

Healthy participants receive cross education training of the elbow flexor (12 rep./set, 3sets, 60%MVC, 180°/s, eccentric).Maximal voluntary contraction, electroencephalogram and electromyogram will record during cross education tasks to determine the effects of cross education training on cortical network and muscle functional connectivity

DETAILED DESCRIPTION:
Cross education (CE) training was observed in 1894, when unilateral strength training of single limb was found to increase in strength of untrained muscle group. CE has potential clinical relevance in rehabilitation for patient who have acute injuries of the limb, post-surgical limb immobilization and certain neurological disorders with unilateral muscle weakness. Although CE has several potential clinical application, the precise physiological mechanisms underlying CE remains unknown. Previous studies reported that CE may involve bilateral cortical activity in both contralateral primary motor cortex (cM1), and ipsilateral primary motor cortex (iM1).In addition, neuroimaging studies have demonstrated that bilateral supplementary motor area, but CE immediate change of functional connectivity in cortical network remains unknown.

The purposes of this study are to investigate the immediate effect of CE training of biceps brachii (1) Immediate change of functional connectivity in cortical network; (2) Immediate change of functional connectivity in cortex and target muscle; (3) Explore immediate change of corticomuscular functional connectivity on maximal voluntary contraction. We hypothesize that (1) Bilateral cortical motor network that exhibit changes in functional connectivity during cross education; (2) Cross education would immediately enhance functional connectivity between cortex and target muscle; (3) Cross education would immediately change corticomuscular functional connectivity on maximal isometric voluntary contraction.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults who are 20-40 years old

Exclusion Criteria:

1. Upper extremity (UE) pain or discomfort
2. Medical condition that substantially influenced their UE strength
3. Experience of UE surgery
4. Paresthesia in UE
5. Open wound on UE

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Corticocortical coherence | Measured immediately after cross education training
  Level of electroencephalography and electromyography synchronization in frequency domain when participants maintain 20% maximal voluntary contraction
Corticomuscular coherence | Measured immediately after cross education training
  Level of electroencephalography and electromyography synchronization in frequency domain when participants maintain 20% maximal voluntary contraction
Maximal voluntary contraction | Measured immediately after cross education training
  The ability to generate maximal voluntary elbow flexor force

CONTACTS AND LOCATIONS:
Overall Officials: Li-Wei Chou, Ph.D., Principal Investigator — Department of Physical Therapy and Assistive and Technology ,National Yang-Ming University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No